CLINICAL TRIAL: NCT01689428
Title: Prospective Randomized Controlled Trail to Assess the Efficacy of EmbryoGen Culture Medium to Improve Ongoing Pregnancy and Implantation Rates in IVF Treatments of Patients With a Previous History of Pregnancy Loss
Brief Title: Ism1 Versus EmbryoGen Media for Embryo Culture in Previous Pregnancy Loss Cases
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Biogenesi (Other)
Responsible Party: Sponsor
Other Study IDs: EG48Asept12; EG1 (Other: Biogenesi Reproductive Medicine Centre)
Record Dates: First submitted 2012-09-10; First posted 2012-09-21 (Estimated); Last update posted 2012-09-21 (Estimated); Status verified 2012-09

CONDITIONS: Infertility; Miscarriage
Keywords: IVF; Embryo culture; Ongoing Pregnancy rate; Ongoing Implantation rate; Miscarriage
MeSH Terms: conditions — Infertility; Abortion, Spontaneous

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- IVF treatment EmbryoGen: Embryo culture in EmbryoGen medium
- IVF treatment ISM1: Embryo culture in ISM1 medium

SUMMARY:
Recently, it has been suggested that culture of embryos in EmbryoGen medium can increase the live birth rate in IVF patients with a previous history of pregnancy loss.

Couples requiring IVF treatment and with a past experience of miscarriage and/or biochemical pregnancy will be included in the study.

Controlled ovarian stimulation protocol will consist of an agonist down regulation and follicular stimulation by recombinant FSH. Fertilization will be achieved by standard IVF or intracytoplasmic sperm injection. Fertilized eggs will be cultured in 6% CO2, 5% O2, 89% N2 atmosphere in microdrops. In the treatment group EmbryoGen culture medium (EG, Origio, Måløv, Denmark) will be adopted throughout the culture period. In the control group, inseminated oocytes will be cultured in standard culture conditions, i.e. IMS1 medium (ISM1, Origio, Måløv, Denmark), maintaining unchanged all other culture conditions.

Procedures of embryo transfer, will be carried out on day 2 using EmbryoGen or ISM1 respectively. The endometrial support will be the same in the two groups.

The investigators will consider ongoing clinical pregnancy as the primary outcome assuming a 25% of increment in ongoing clinical pregnancy rate in the group with EmbryoGen medium. As secondary outcome the investigators will assume a 5% of increment in ongoing implantation rate after 12 weeks in the group with EmbryoGen medium.

ELIGIBILITY:
Inclusion Criteria:

- At least one (maximum 3) miscarriage and/or biochemical pregnancy after ART treatment

Exclusion Criteria:

* Frozen spermatozoa
* Frozen oocytes
* women with PCO and PCOS
* women with more than 4 ART treatments

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Infertile couple with an indication for standard IVF or intracytoplasmic sperm injection. Moreover all couples had at least a previous miscarriage and/or biochemical pregnancy experience after ART treatment.
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2012-09; Primary Completion 2013-06 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Ongoing Pregnancy Rate after 12 weeks of gestation | 12 weeks after conception

SECONDARY OUTCOMES:
Ongoing Implantation Rate after 12 weeks of gestation | 12 weeks after conception

CONTACTS AND LOCATIONS:
Overall Officials: Mariabeatrice Dal Canto, PhD, Principal Investigator — Biogenesi Reproductive medicine Centre
Locations (1):
- Biogenesi Reproductive Medicine Centre, Monza, MB, Italy

REFERENCES:
- [Background] Agerholm I, Loft A, Hald F, Lemmen JG, Munding B, Sorensen PD, Ziebe S. Culture of human oocytes with granulocyte-macrophage colony-stimulating factor has no effect on embryonic chromosomal constitution. Reprod Biomed Online. 2010 Apr;20(4):477-84. doi: 10.1016/j.rbmo.2009.12.026. Epub 2009 Dec 28. PMID 20129825